CLINICAL TRIAL: NCT06771557
Title: Evaluation of Usage and Efficacy of the 656 Online Platform for Reducing Caregiver Stress in Chinese Caregivers: Longitudinal Open-trial Study
Brief Title: Evaluation of Usage and Efficacy of the 656 Online Platform for Reducing Caregiver Stress in Chinese Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Wendy Zhang Wen, Assistant Professor, Hong Kong Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2021-39-E
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stoke; Dementia; Fall and Fractures Prevention
Keywords: Online Platform; Caregivers; Caregiver stress
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: A longitudinal open-trial study design was applied (N=287) with outcome measures administered at baseline, 3-month follow-up, and 15-month follow-up. Primary outcomes included changes in caregiver stress, caregiver preparedness, and competence. The user profile was explored by comparing the characteristics of participants in user group and non-user group. User satisfaction and engagement were also reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Users of the 656 Online Platform (Experimental): The experimental arm includes caregivers of the elderly with three targeted disorders (stroke, dementia, and fall-related fractures) who used the 656 Online Platform. The 656 Platform provides valuable information regarding three common ailments among the elderly, namely stroke, dementia, and fall-related fractures.
  Interventions: Other: 656 Online Platform
- Non-users of the 656 Online Platform (No Intervention): This arm includes caregivers of the elderly with three targeted disorders (stroke, dementia, and fall-related fractures) who did not use the 656 Online Platform. The 656 Platform provides valuable information regarding three common ailments among the elderly, namely stroke, dementia, and fall-related fractures.

INTERVENTIONS:
Other: 656 Online Platform — The 656 Platform provides valuable information regarding three common ailments among the elderly, namely stroke, dementia, and fall-related fractures. Serving as an online platform, the 656 Platform incorporates a Chatbot feature that facilitates connections between local caregivers, social workers, and community members to various services. Serving as an online platform, the 656 Platform incorporates an AI Chatbot and a Live Chat feature that facilitates connections between local caregivers, social workers, and community members to various services. Apart from this, the 656 Platform offers several features that enhance its functionality and user experience, including problem-based elderly resource database, interim care solutions, exchange forum, data analytics and research, and professional knowledge and resources.
  Arms: Users of the 656 Online Platform

SUMMARY:
This study aimed to assess the efficacy of a new online platform, 656 Online Platform, in Hong Kong in reducing caregiver stress and enhancing caregiver preparedness and competence of caring for older adults with stroke, dementia, and fracture, investigate the factors influencing the usage of the online platform, and examine user satisfaction and engagement.

DETAILED DESCRIPTION:
The informal caregivers of older adults with serious health problems, especially for stroke, dementia, and fracture, are facing numerous caregiving stress. The online platform can be a cost-effective way to support caregivers and reduce their caregiving stress.

A new online platform, the 655 Online Platform, was developed by St. James Settlement in Hong Kong, to provide caregivers with appropriate information and support, attempting to reduce their pressure. Therefore, this study was launched to evaluate the efficacy of a new online platform in reducing caregiver stress and enhancing caregiver preparedness and competence in caring for older adults with stroke, dementia, and fracture, investigate the factors influencing the usage of the online platform, and examine user satisfaction and engagement.

A longitudinal open-trial study design was applied (N=287) with outcome measures administered at baseline, 3-month follow-up, and 15-month follow-up. Primary outcomes included changes in caregiver stress, caregiver preparedness, and competence. The user profile was explored by comparing the characteristics of participants in user group and non-user group. User satisfaction and engagement were also reported.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers who are Chinese citizens aged 18 or above and provide care for elderly individuals aged 65 or above diagnosed with stroke, dementia, or fall-related fractures

Exclusion Criteria:

* Family caregivers who have been diagnosed with severe mental or physical illness or have impairments in cognitive function, such as comprehension, memory, observation, and other related abilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Caregiver stress | From the baseline survey to the second follow-up survey at 15 months
  Caregiver stress was measured by Modified Caregiver Strain Index (C-M-CSI). It consists of 13 items with a total score ranging from 0 to 26. Each item is rated by a score of 0 (no), 1 (yes, sometimes) or 2 (yes, always). A higher score suggests a higher amount of strain felt by caregivers. The C-M-CSI demonstrated good psychometric properties in the Chinese population.
Preparedness for caregiving | From the baseline survey to the second follow-up survey at 15 months
  Preparedness for caregiving was measured by the Chinese version of Preparedness for Caregiving Scale. The scale consists of 8 items that ask careers how well prepared they believe they are for multiple domains of caregiving. Each item is rated by a five-point Likert scale from 0 (not at all prepared) to 4 (very well prepared) with a total score from 0 to 32. The scale showed good reliability and validity in the Chinese population.
Caregiver competence | From the baseline survey to the second follow-up survey at 15 months
  Caregiver competence was measured by the Chinese version of Caregiver Competence Scale (CCS-C).The scale includes 4 items to assess the sufficiency of a caregiver's performance as administered by the caregiver. A higher score indicates a better sense of competence. The CCS-C demonstrated good psychometric properties in the Chinese caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Ha WONG, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The privacy and personal information of the respondents are highly valued and strictly protected.